CLINICAL TRIAL: NCT00992147
Title: A Phase II/III Clinical Study of ANTG-adip for the Treatment of Depressed Scar to Evaluate Safety and Efficacy
Brief Title: Safety and Efficacy of Autologous Cultured Adipocytes in Patient With Depressed Scar
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Anterogen Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANTG-adip-301
Record Dates: First submitted 2009-09-28; First posted 2009-10-09 (Estimated); Last update posted 2009-10-09 (Estimated); Status verified 2009-10

CONDITIONS: Depressed Scar

ARMS (1):
- autologous cultured adipocytes (Experimental)
  Interventions: Drug: Adipocell

INTERVENTIONS:
Drug: Adipocell — autologous cultured adipocytes (ANTG-adip)

SUMMARY:
Autologous cultured adipocytes (ANTG-adip) is produced by well-established techniques including cell harvesting from lipoaspirates, expansion of adipose tissue derived stem cells, and differentiation into pure and immature adipocytes. This was an open-label, dose-escalation study. Patients are given subcutaneous injection of ANTG-adip and followed for 12 weeks according to the clinical trial protocol.

ELIGIBILITY:
Inclusion Criteria:

* older than 19 years
* depressed scar less than volume of 5 ml
* negative for urine beta-HCG for women of childbearing age
* agreement to participate, with signed informed-consent

Exclusion Criteria:

* failure to meet inclusion criteria
* any immune-suppressive drug, corticosteroid or cytotoxic drug within the previous 30 days
* allergy to bovine-derived materials
* Diagnosis of cancer, AIDS, HBV or HCV.
* Patient has a lot of hairs or a tattoo on depressed site
* Insufficient adipose tissue for manufacturing of ANTG-adip
* Patient has depressed scar caused by a malignant tumor
* Patient whom investigator consider is not suitable in this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2004-05; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Efficacy: recovery rate(%) | week 12
Safety: clinically measured abnormality of laboratory tests and adverse events, Injection site observation, Immune rejection test

SECONDARY OUTCOMES:
Recovery rate (%) | day 7, 14, 21, 28 days and week 8
A digital photograph | day 1, 3, 7, 14, 21, 28, week 8 and week 12
Patient satisfaction | week 12

CONTACTS AND LOCATIONS:
Overall Officials: Gab-sung Oh, M.D, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea